CLINICAL TRIAL: NCT02402582
Title: Family-Centered Empowerment Model With Four-stage Including Perceived Threat With Group Discussion Method, Self-efficacy With Problem Solving Method, Self-esteem With Educational Partnership, and Outcome and Process Evaluations
Brief Title: Effect of Family-Centered Empowerment Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Tarbiat Modarres University (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, Baqiyatallah Medical Sciences University, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BMSU
Record Dates: First submitted 2015-03-20; First posted 2015-03-30 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Acute Myocardial Infarction: Rehabilitation Phase
Keywords: Family-Centered Empowerment Model; Quality of life; Perceived stress; Anxiety; Myocardial infarction; Clinical trial; Iran
MeSH Terms: conditions — Anxiety Disorders; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: All patients had similar inpatient rehabilitation programs. Both groups exercised for 0-2h/day. Walking distance was measured using a Fitbit (Fitbit, San Francisco, USA). Routine care included education on smoking cessation and education on food selection.
  FCEM: Daily exercise occurred between 8-10 AM and was supervised by designated family members. Investigators randomly attended sessions in an unannounced fashion. Physical therapy consultation was available on investigator request. Exercise data were independently collected from the patient and their designated family member on a weekly basis (κ statistic=0.9).
  Control: Patients exercised daily, at any time. Sessions were supervised by family members. Investigators did not attend sessions. Exercise data were independently collected from the patient and their designated family member on a weekly basis (κ statistic=0.4).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family-Centered Empowerment Model (Experimental): Have the same in-patient, pre-intervention, and post-intervention follow-up care as Control Group. However, rather than routine care and follow-up during the intervention period, they recieved than 4 stage intervention using the Family Centered Empowerment Model.
  Interventions: Other: Family-centered empowerment model
- Control (Active Comparator): Same in-patient, pre-intervention, and post-intervention follow-up care as Experimental Group. However, rather than 4 stage intervention they receive routine care and follow-up.
  Interventions: Other: Control

INTERVENTIONS:
Other: Family-centered empowerment model — FCEM and Control groups had similar inpatient care. Patients in the intervention group received care employing the FCEM in four stages. Stage 1: Awareness and cognition. During 3-5 group sessions they were evaluated for their insight into their perceived illness severity and perceived sensitivity, or the degree to which they felt threatened by their illness. Stage 2: Expectations. 3-5 sessions. Stage 3: Acceptance. Assessed using an educational participation method in group discussion. Stage 4: Formative summative evaluations. The formative evaluation encourages patients to internalize their locus of control by seeing his/her self-empowerment (increasing self-responsibility about their health). Summative evaluations were performed to evaluate the influence of the intervention on HRQoL dimensions, perceived stress and anxiety -- assessed at baseline and at 3 months post-intervention. Empowerment was measured at baseline and at 10 days post-intervention by deploying FCEM questionnaires.
  Other Names: FCEM
  Arms: Family-Centered Empowerment Model
Other: Control — FCEM and Control groups had similar inpatient care. Upon discharge the Control group underwent routine care and follow-up.
  Arms: Control

SUMMARY:
The objective of this study was to evaluate the effectiveness of a FCEM-focused hybrid CR program for survivors of myocardial infarction (MI). The study sought to compare the long-term impact of FCEM-based intervention with a standard CR program in terms of mortality rates and different aspects of health related quality of life (HRQoL), which includes soft outcomes such as levels of stress, anxiety, psychological distress, quality of life (QoL), and hard outcomes such as the percentage of ejection fraction (EF), independent functioning, and functional exercise capacity status.

DETAILED DESCRIPTION:
The investigators conducted a triple-blind randomized controlled clinical trial study in patients admitted for MI to the CCU of an academic teaching hospital from June 2012 to January 2023. The study was approved by the institutional investigative review board at Tarbiat Modares University and Baqiyatallah University of Medical Sciences. Patients were block randomized to receive either standard home cardiac rehabilitation (CR) or CR using the Family-centered Empowerment Model (FCEM) strategy. Patients had not previously gone through CR programs. The difference between the two groups was not disclosed at any point. Patients consented knowing that they would receive cardiac rehabilitation, but without knowing the details. Patients and their designated family/friend were enrolled as a 'unit'. Patient empowerment was measured with FCEM questionnaires pre-intervention and post-intervention for a total of 9 assessments. Quality-of-life, perceived stress, state and trait anxiety, psychological distress, independent functioning, and functional exercise capacity status were assessed using the 36-Item Short Form Health Survey (SF-36), the 14-item Perceived Stress, the 20-item State and 20-item Trait Anxiety questionnaires, Kessler Psychological Distress Scale,Barthel Index (BI) activities of daily living index, six-minute walk test (6MWT), and free walking index (FWI), respectively. In addition, echocardiography was used to measure ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Being within the age-range of 45 to 85 years old
* having the minimum literacy for reading and writing
* being hospitalized due to MI for the first time
* verification of MI by clinical symptoms
* enzyme-serum tests and cardiograph changes
* lack of participation in the any related educational course simultaneously with the execution of intervention
* patients' willingness toward participating in the research
* having no psychological problems
* ability to fill out the questionnaire and participating in the empowerment program.

Exclusion Criteria:

* any offending items from mentioned criteria.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 10-year
  5-year, 7-year, and 10-year mortality rates of MI survivors who received a FCEM-focused hybrid CR program as intervention group compared with those who received a standard CR program as control group

SECONDARY OUTCOMES:
Patient Stress | 48 months
  14-item Perceived Stress Questionnaire (PSQ-14)
Anxiety | 48 months
  Beck 20-Item state and 20-Item trait anxiety Questionnaires
Level of quality of life | 48 months
  the 36-Item Short Form Health Survey (SF-36)
psychological distress | 48 months
  Psychological Distress Scale (K10)

OTHER OUTCOMES:
Ejection Fraction | 48 months
  Measured by trans-thoracic echocardiography
Independent functioning | 48 months
  Barthel Index (BI) activities of daily living index
Functional exercise capacity status | 48 months
  six-minute walk test (6MWT), and free walking index (FWI)

CONTACTS AND LOCATIONS:
Overall Officials: Amir vahedian-azimi, Resea fellow, Principal Investigator — BMSU

REFERENCES:
- [Result] Vahedian-Azimi A, Miller AC, Hajiesmaieli M, Kangasniemi M, Alhani F, Jelvehmoghaddam H, Fathi M, Farzanegan B, Ardehali SH, Hatamian S, Gahremani M, Mosavinasab SM, Rostami Z, Madani SJ, Izadi M. Cardiac rehabilitation using the Family-Centered Empowerment Model versus home-based cardiac rehabilitation in patients with myocardial infarction: a randomised controlled trial. Open Heart. 2016 Apr 19;3(1):e000349. doi: 10.1136/openhrt-2015-000349. eCollection 2016. PMID 27110376
- [Derived] Vahedian-Azimi A, Sanjari MJ, Rahimi-Bashar F, Gohari-Mogadam K, Ouahrani A, Mustafa EMM, Ait Hssain A, Sahebkar A. Cardiac Rehabilitation Using the Family-Centered Empowerment Model is Effective in Improving Long-term Mortality in Patients with Myocardial Infarction: A 10-year Follow-Up Randomized Clinical Trial. High Blood Press Cardiovasc Prev. 2024 Mar;31(2):189-204. doi: 10.1007/s40292-024-00636-2. Epub 2024 Apr 2. PMID 38564167
- See also: "Open Heart" site for full text — http://openheart.bmj.com/content/3/1/e000349